CLINICAL TRIAL: NCT04532502
Title: Work Environment's Impact on the Sex Ratio of the Children of Resuscitation Anesthesia Assistants
Brief Title: Impact of Anesthetic Environment the Sex Ratio of the Children of Female Assistants
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Professor, University of Liege
Other Study IDs: GENREANES
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Anesthesia, General; Anesthetics Adverse Reaction
Keywords: Anesthesia care providers; offspring sex ratio; Inhalation induction of anesthesia
MeSH Terms: interventions — Anesthetics, Inhalation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: All female assistants in anesthesia
  Interventions: Drug: Anesthetics, Inhalation

INTERVENTIONS:
Drug: Anesthetics, Inhalation — Work environmental exposure

SUMMARY:
The aims of this multi center retrospective study was to determine:

* whether the sex ratio of the offspring of female assistants in anesthesia-resuscitation differs from that of the population at large
* whether the assistants' work environment at the time of their offspring's conception influences the sex of their offspring

ELIGIBILITY:
Inclusion Criteria:

* Female assistants in anesthesia-resuscitation in the Wallonia-Brussels Federation (Belgium) who conceived one or more children in the course of their training between 2009 and 2019 and who delivered before the end of 2019 (cut-off: midnight on 31 December 2019)

Exclusion Criteria:

* Male assistants in anesthesia-resuscitation
* Female assistants in anesthesia-resuscitation who trained before 2009 or after 2019.
* Female assistants in anesthesia-resuscitation who relied on medically assisted reproduction.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The anesthesia department of the three French-speaking universities in Belgium wimp e-mail a questionnaire to all female assistants in anesthesia-resuscitation via a system similar to Survey Monkey. The data will be completely anonymized through those of such a system.
  Reminder will be e-mailed 1 and 3 months after the questionnaire is sent out. Filling the questionnaire will be equated with consent
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Offspring sex ratio | 5 years (duration of anesthesia training)
  Offspring sex ratio of female anesthesia assistants will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Philippe J Van der Linden, MD, Study Director — CHU Brugmann, Free University of Brussels, Belgium
Locations (1):
- ULiege, Liège, Belgium

REFERENCES:
- [Background] Gupta D, Kaminski E, McKelvey G, Wang H. Firstborn offspring sex ratio is skewed towards female offspring in anesthesia care providers: A questionnaire-based nationwide study from United States. J Anaesthesiol Clin Pharmacol. 2013 Apr;29(2):221-7. doi: 10.4103/0970-9185.111728. PMID 23878446
- [Background] Leroy C, Daelemans C, Debauche C, Van Leeuw V. Santé périnatale en Wallonie - année 2017, Centre d'Epidémiologie Périnatale 2019.